CLINICAL TRIAL: NCT02796404
Title: Effectiveness of a Homebased Cardiac Rehabilitation Program of Mixed Surveillance Using NUUBO Monitoring Vest in Patients With Ischemic Heart Disease at Moderate Cardiovascular Risk
Brief Title: Homebased Monitoring Cardiac Rehabilitation Program
Acronym: NUUBO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUUBO
Record Dates: First submitted 2016-05-23; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Homebased Cardiac Rehabilitation Program After Ischemic Heart Disease
Keywords: home monitoring; cardiac monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homebased cardiac rehabilitation program (Experimental): Homebased Cardiac rehabilitation program with monitoring vest and mixed surveillance.
  Interventions: Device: Homebased cardiac rehabilitation program; Other: Traditional cardiac rehabilitation program
- Traditional cardiac rehabilitation (Other): Multidisciplinary program in a cardiac rehabilitation gym. Routine clinical practice
  Interventions: Other: Traditional cardiac rehabilitation program

INTERVENTIONS:
Device: Homebased cardiac rehabilitation program — homebased cardiac rehabilitation program with monitoring vest Nuubo
  Arms: Homebased cardiac rehabilitation program
Other: Traditional cardiac rehabilitation program — multidisciplinary intervention in cardiac rehabilitation gym

SUMMARY:
The current state of mobile communication and technology is a tool to support home programs for chronic disease management, useful to facilitate access to these types of programs, because the investigators could obtain telematics information about the parameters, reducing cardiovascular risk factors and cardiovascular morbidity and mortality.

DETAILED DESCRIPTION:
The current state of mobile communication and technology is a tool to support home programs for chronic disease management, useful to facilitate access to these types of programs, because the investigators could obtain telematics information about the parameters, reducing cardiovascular risk factors and cardiovascular morbidity and mortality.

Once the patient qualifies for inclusion in the study and has signed informed consent it is included in a list where randomized 7 patients in the experimental group (home-based cardiac rehabilitation Nuubo monitoring vest) and 7 patients are assigned to traditional cardiac rehabilitation group.

ELIGIBILITY:
Inclusion Criteria:

All of them:

* Age ≤ 80 years.
* Stable Ischemic heart disease, revascularized by angioplasty or underwent surgery by coronary bypass <= one year from the acute episode.
* Good cognitive level.
* Ability to perform aerobic exercise tape or cycle ergometer.
* Understand the use of a mobile Smartphone or Tablet.
* Signature of informed consent.

And at least one of the following:

* Ventricular dysfunction by Ejection Fraction (FE) 40 - 50%.
* Functional capacity 5-7 metabolic equivalents (METS).
* Raising the blood pressure with the effort.

Exclusion Criteria:

* Presence of malignant arrhythmias such as ventricular fibrillation outside the acute phase of Acute myocardial infarction (AMI) (> 24 h after AMI), ventricular tachycardia, Atrioventricular block of 2nd degree and 3rd degree, Atrial fibrilation (FA) in patients with Wolf Parkinson White, fibrillation or paroxysmal atrial flutter with response ventricular quickly and hemodynamic deterioration, premature ventricular contractions increases during exertion, paroxysmal supraventricular tachycardia uncontrolled.
* Previous infarcts.
* Hypotensive response to exercise.
* Myocardial Ischemia valued at exercise test.
* Unstable Angina.
* Nonrevascularizable disease.
* Poorly controlled hypertension baseline.
* Killip III and IV Killip.
* No collaborator.
* Valvular heart disease associated.
* Pacemaker or Implantable Cardioverter Defibrillator.
* Pathology of musculoskeletal, neurological or breathing that impair the ability of prolonged ambulation.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness measured by exercise testing and control of cardiovascular risk factors | During 12 months
  functional capacity obtained by exercise testing and control of cardiovascular risk factors.

SECONDARY OUTCOMES:
Results of homebased cardiac rehabilitation monitoring a traditional cardiac rehabilitation program | During 12 months
  comparing the results of functional capacity measured by exercise testing and control of cardiovascular risk factors between the two groups
Adherence to these programs | 3, 6 and 12 months
  see adherence to these program at 3, 6 months and a year depending on the habit of exercise and control of cardiovascular risk factors.
Safety to these program | During 12 months
  See the safety of home cardiac rehabilitation program of mixed surveillance compared to traditional cardiac rehabilitation program to checking the existence of adverse cardiac events.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Bravo, MD, Principal Investigator — rbravoescobar@yahoo.es
Locations (3):
- Spain (3):
  - Hospital Mediterráneo, Almería, Almería
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Z, Jia X, Li J, Mei Z, Yang L, Yan C, Han Y. Efficacy and Safety of Hybrid Comprehensive Telerehabilitation (HCTR) for Cardiac Rehabilitation in Patients with Cardiovascular Disease: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Occup Ther Int. 2023 Aug 9;2023:5147805. doi: 10.1155/2023/5147805. eCollection 2023. PMID 37593110
- [Derived] Bravo-Escobar R, Gonzalez-Represas A, Gomez-Gonzalez AM, Heredia-Torres A. Effectiveness of e-Health cardiac rehabilitation program on quality of life associated with symptoms of anxiety and depression in moderate-risk patients. Sci Rep. 2021 Feb 12;11(1):3760. doi: 10.1038/s41598-021-83231-y. PMID 33580174
- [Derived] Bravo-Escobar R, Gonzalez-Represas A, Gomez-Gonzalez AM, Montiel-Trujillo A, Aguilar-Jimenez R, Carrasco-Ruiz R, Salinas-Sanchez P. Effectiveness and safety of a home-based cardiac rehabilitation programme of mixed surveillance in patients with ischemic heart disease at moderate cardiovascular risk: A randomised, controlled clinical trial. BMC Cardiovasc Disord. 2017 Feb 20;17(1):66. doi: 10.1186/s12872-017-0499-0. PMID 28219338